CLINICAL TRIAL: NCT00381108
Title: A Randomized, Double Blinded, Controlled Clinical Trial of Pomegranate Tablets vs Placebo: Effects on Symptoms of Benign Prostatic Hyperplasia
Brief Title: Study of the Effects of Pomegranate Tablets on Enlarged Prostates
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Irvine (Other)
Collaborators: Pomegranate Health (Industry); Jarrow Pharmaceuticals (Unknown)
Responsible Party: Leland Ronningnen, MD, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-4373
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomegranate Tablet (Experimental)
  Interventions: Drug: Pomegranate Tablet
- Placebo Tablet (Placebo Comparator)
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Placebo Tablet — Two tablets, twice daily.
  Arms: Placebo Tablet
Drug: Pomegranate Tablet — Two tablets, twice daily.
  Arms: Pomegranate Tablet

SUMMARY:
To determine whether pomegranate tablets have a therapeutic effect on Benign Prostatic Hyperplasia.

DETAILED DESCRIPTION:
Patients with newly diagnosed benign prostatic hyperplasia (BPH) will be recruited from the urology clinic at UCI medical center for this study as indicated in section 4. Once recruited, patients will be randomized into two groups - placebo and pomegranate tablets.

Prior to randomization, there will be a 6 week run-in period in which the basal parameters will be established. The basal parameters include a complete history and physical exam including an AUA symptom questionnaire and men's sexual health questionnaire, urine culture, urinalysis, PSA, serum chemistry (sodium, potassium, chloride, bicarbonate, BUN, creatinine, glucose), serum free testosterone, serum dihydrotestosterone, maximum urinary flow rate (Qmax), post void residual bladder volume, and prostate volume measurement via Trans-rectal ultrasound. Then patients will be randomized either to the study group or to the control group using a random number generator. All of the study subjects will be counseled to take one capsule daily in the morning and not to consume any other prostate supplements, or other forms of medical or herbal therapy for BPH.

Patients will be asked to come in every 2 months for the following tests and questionnaires to be administered:

1. AUA Symptoms Score sheet
2. Men's Sexual Health Questionnaire
3. Urine culture
4. Urinalysis
5. PSA
6. Serum chemistry (sodium, potassium, chloride, bicarbonate, BUN, creatinine, glucose)
7. Serum free testosterone
8. Serum 5-dihydrotestosterone
9. Maximum urinary flow rate (Qmax)
10. Post void residual check
11. Prostate volume measurement via Trans-rectal ultrasound

Maximum blood volume that will be drawn for each blood draw is 10 ml (2 table spoon), and the maximum blood draws per patient is 3 per person if there is no crossover and 6 if there is a crossover. Prior to all blood draw, patients will be asked to refrain from sexual intercourse for at least 48 hrs.

Patients with severe BPH (AUA symptom score 20 and above) or those already on other forms of medical therapy such as prescription finasteride, terazosin, or tamsulosin, propecia (for hair loss) or have any history of prostate surgery are not eligible to participate in this study. Also, patients who are taking non prescription supplements such as Saw Palmetto, B-sitosterol, vitamin E, quercetin, will not be included in the study. One group (n = 10) will take the pomegranate tablet. Group 2 (n = 10) will take 1 placebo tablet in the morning daily. Both pomegranate tablets and placebo will be provided by the Pomegranate Health Company.

Prior to randomization, there will be a 6-week run-in time because voiding parameters are notoriously variable. During this run-in time, patients will be asked to return to clinic every two weeks to measure maximum urinary flow and post-void residual bladder volume.

After a six-month period, each subject will be crossed over individually from placebo to active treatment, and from active treatment to placebo. The total anticipated timeline for the study is 12 months.

If early termination from the study is requested a final evaluation will be given. The final evaluation of the study will entail a standard office visit with blood collection and final AUA symptoms score and Men's sexual health questionnaire, and a transrectal ultrasound of the prostate measuring the same parameters as in the previous office visits. Subsequently, recommendations will be made by a urologist regarding the standard treatment options for BPH.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinically diagnosed with mild to moderate BPH (AUA symptom score <20)

Exclusion Criteria:

* Patient with severe BPH (AUA symptom score >21)
* Currently using any other forms of medical therapy, prescription finasteride, terazosin, tamsulosin or propecia (for hair loss).
* Prior Transurethral resection of the prostate (TURP).
* Using non-prescription supplements such as Saw Palmetto, B-sitosterol, vitamin E, and quercetin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Patients w/ BPH symptoms will be followed w/ AUA symptom questionnaires & exams; in addition, urinary flow rate & post void residual checks will be done to determine whether patients on pomegranate tablets have a reduction in symptoms. | Time points in which data is collected are initial visit, two weeks, four weeks, and 2, 4, 6, 8, 10, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Ronningen, MD, Principal Investigator — UCIMC Department of Urology
Locations (2):
- United States (2):
  - VA Long Beach, Long Beach, California
  - University of California, Irvine-Department of Urology, Orange, California